CLINICAL TRIAL: NCT00237770
Title: Prevention of Low Blood Pressure in Persons With Tetraplegia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3600-R
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Hypotension; Spinal Cord Injury
Keywords: Blood Pressure; Cardiovascular Autonomic Control; Nitric Oxide; NOS Inhibitor; Orthostatic Hypotension; Spinal Cord Injury; Tetraplegia
MeSH Terms: conditions — Hypotension; Spinal Cord Injuries; Hypotension, Orthostatic; Quadriplegia | interventions — NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Placebo Comparator): Placebo control (normal saline) is employed on a separate visit during procedure.
  Interventions: Drug: N-Nitro L-arginine-methylester (L-NAME); Procedure: Head-up Tilt maneuver

INTERVENTIONS:
Drug: N-Nitro L-arginine-methylester (L-NAME) — A non-specific inhibitor of the nitric oxide synthase enzyme.
Procedure: Head-up Tilt maneuver — Participant will be placed onto tilt table and brought to 15 degrees of head up tilt for 60 minutes (intravenous infusion time). After this time, a progressive increase to 45 degrees will be completed with a 10 degree increase every 5 minutes. Participant will remain at 45 degrees for 45 minutes or until symptom onset.

SUMMARY:
The aim of this investigation is to determine the blood pressure response to NOS inhibition, with L-NAME, in persons with tetraplegia compared to non-SCI control subjects and to establish if blood pressure can be increased while upright in those with tetraplegia. If blood pressure is increased with NOS inhibition in persons with tetraplegia, this would improve our treatment of the condition of low blood pressure during seated postures in individuals with tetraplegia.

DETAILED DESCRIPTION:
Despite disruption of central command of the vasculature during orthostatic maneuvers, individuals with tetraplegia are generally able to be seated in an upright position for long periods of time without developing symptoms of orthostatic intolerance. It must be appreciated however, that orthostatic hypotension may occur unpredictably in persons with chronic tetraplegia. This may result in a range of symptoms due to cerebral hypoperfusion from mild reduction in mental acuity to loss of consciousness. Nitric oxide (NO) is the most potent endogenous vasodilator which is synthesized by the enzyme NO synthase (NOS) and may be largely responsible for orthostatic hypotension in individuals with immobilizing conditions. Recent evidence suggests an up-regulation of inducible nitric oxide synthases (NOS) activity with prolonged exposure to hind limb suspension. The effects of NOS inhibition during orthostasis on blood pressure regulation in those with chronic tetraplegia may provide insight into effective pharmacological therapy to reduce or prevent pathologic orthostatic changes. Treatment with a NOS inhibitor may facilitate the process of mobilization in those with acute higher cord lesions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year olds.
* Non-ambulatory Chronic tetraplegia (1 year after acute SCI).

Exclusion Criteria:

* central nervous system disease (other than SCI) e.g., multiple sclerosis, amyotrophic lateral sclerosis, syringomyelia, tabes dorsalis;
* peripheral neuropathies;
* surgical sympathectomy;
* coronary heart and/or artery disease;
* anemia;
* hypertension;
* renal function abnormalities;
* diabetes mellitus;
* pituitary insufficiency;
* adrenal insufficiency;
* hypothyroidism; and
* medications known to affect the cardiovascular system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Wecht JM, Weir JP, Krothe AH, Spungen AM, Bauman WA. Normalization of supine blood pressure after nitric oxide synthase inhibition in persons with tetraplegia. J Spinal Cord Med. 2007;30(1):5-9. doi: 10.1080/10790268.2007.11753907. PMID 17385265
- [Result] Wecht JM, Weir JP, Goldstein DS, Krothe-Petroff A, Spungen AM, Holmes C, Bauman WA. Direct and reflexive effects of nitric oxide synthase inhibition on blood pressure. Am J Physiol Heart Circ Physiol. 2008 Jan;294(1):H190-7. doi: 10.1152/ajpheart.00366.2007. Epub 2007 Oct 26. PMID 17965289
- [Result] Wecht JM, Radulovic M, Lafountaine MF, Rosado-Rivera D, Zhang RL, Bauman WA. Orthostatic responses to nitric oxide synthase inhibition in persons with tetraplegia. Arch Phys Med Rehabil. 2009 Aug;90(8):1428-34. doi: 10.1016/j.apmr.2009.02.004. PMID 19651280
- [Result] Wecht JM, Radulovic M, Rosado-Rivera D, Zhang RL, LaFountaine MF, Bauman WA. Orthostatic effects of midodrine versus L-NAME on cerebral blood flow and the renin-angiotensin-aldosterone system in tetraplegia. Arch Phys Med Rehabil. 2011 Nov;92(11):1789-95. doi: 10.1016/j.apmr.2011.03.022. Epub 2011 Jul 16. PMID 21762873
- [Derived] La Fountaine MF, Wecht JM, Bauman WA. Acute nitric oxide synthase inhibition and cardiac conduction in persons with spinal cord injury: a short report. Pharmazie. 2013 Apr;68(4):245-50. PMID 23700789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured from January 2006 through May 2009; participants were recruited from the James J Peters VA Medical Center and the surrounding community.
Pre-assignment Details: No subject was excluded after enrollment prior to participation.
Groups:
- Tetraplegic Subjects: All tetraplegic subjects underwent a head-up tilt maneuver to determine systolic blood pressure responses to placebo L-NAME 1.0 mg/kg and L-NAME 2.0 mg/kg. Subjects with tetraplegia visited the laboratory on 3 separate occasions.
- Control Subjects: Systolic blood pressure responses to head-up tilt were determined in non-spinal cord injured control subjects following placebo administration. Control subjects visited the laboratory for 1 visit.
Period: Overall Study
Arm/Group | Tetraplegic Subjects | Control Subjects
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Individuals With Tetraplegia: Systolic blood pressure responses to head-up tilt were determined after placebo, L-NAME (1.0 mg/kg) and L-NAME administration (2.0 mg/kg) administration.
- Able-bodied Controls: Systolic blood pressure responses to head-up tilt were determined in able-bodied controls following placebo administration
- Total: Total of all reporting groups
Arm/Group | Individuals With Tetraplegia | Able-bodied Controls | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10) | 33 (9) | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure During Head-up Tilt
Description: Average systolic blood pressure over 45 minutes at 45 degrees of head-up tilt.
Time Frame: Average systolic blood pressure during head-up tilt (45 degrees) comparing active drug (L-NAME: 1.0 and 2.0 mg/kg) to placebo.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Tetraplegic Systolic Blood Pressure Responses to Placebo: Systolic blood pressure responses to head-up tilt were determined after placebo administration in persons with tetraplegia
- Control Systolic Blood Pressure Responses to Placebo: Systolic blood pressure responses to head-up tilt were determined in non spinal cord injured controls following placebo administration
- Tetraplegic Systolic Blood Pressure Responses to L-NAME 1.0 mg: Systolic blood pressure responses to head-up tilt were determined following administration of L-NAME (1.0 mg/kg)
- Tetraplegic Systolic Blood Pressure Responses to L-NAME 2.0 mg: Systolic blood pressure responses during head-up tilt were determined following L-NAME administration (2.0 mg/kg)
Arm/Group | Tetraplegic Systolic Blood Pressure Responses to Placebo | Control Systolic Blood Pressure Responses to Placebo | Tetraplegic Systolic Blood Pressure Responses to L-NAME 1.0 mg | Tetraplegic Systolic Blood Pressure Responses to L-NAME 2.0 mg
Number analyzed (Participants) | 9 | 7 | 9 | 9
mmHg | 91.80 (20.96) | 108.10 (12.18) | 112.04 (28.01) | 129.94 (26.43)

ADVERSE EVENTS:
Arm/Group | Tetraplegic Systolic Blood Pressure Responses to Placebo | Control Systolic Blood Pressure Responses to Placebo | Tetraplegic Systolic Blood Pressure Responses to L-NAME 1.0 mg | Tetraplegic Systolic Blood Pressure Responses to L-NAME 2.0 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
The small sample of subjects tested and the heterogeneity of spinal lesions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No